CLINICAL TRIAL: NCT02935647
Title: Burst Suppression Anesthesia for Treatment of Severe Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brian Mickey, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00090838
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Experimental): Participants will receive intravenous propofol titrated rapidly at 100-200 mcg/kg/min to reach 80% burst-suppression and then maintained there for 15 minutes, after which propofol administration will be discontinued and the participant will be allowed to awaken.
  Interventions: Drug: Diprivan

INTERVENTIONS:
Drug: Diprivan
  Other Names: Propofol

SUMMARY:
This study is designed to determine if the antidepressant effects of deep anesthesia via propofol are related to EEG burst suppression.

DETAILED DESCRIPTION:
Ten individuals with treatment resistant major depressive disorder will undergo 10 treatments of deep anesthesia via propofol over a 3-week period. Depression will be evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of Major Depressive Disorder (MDD) or bipolar Disorder (I or II, most recent episode must be depression

  * Failed at least 2 anti-depressant treatments and no ECT in past 6 months
  * Age between 18-55 years
  * BMI < 35
  * Hamilton Rating Scale for Depression (HSRD) score > 18
  * Quick Inventory of Depression Scale (QIDS) score > 10.

Exclusion Criteria:

* • Diagnosis of primary psychotic disorder, dysthymia, or personality disorder

  * Significant pre-morbid cognitive impairment
  * Hypertension and current use of ACE inhibitor or AR blocker medications
  * Symptomatic coronary artery disease or congestive heart failure
  * History of transient ischemic or neurologic signs during the past year
  * History of or susceptibility to malignant hyperthermia
  * Contraindication to isoflurane or propofol anesthesia (as determined by anesthesiologist)
  * Diabetes requiring insulin
  * Poor kidney function
  * Chronic use of benzodiazepines or opioids
  * Individuals incompetent to provide consent (e.g. catatonic, psychotic).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 3 weeks

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Neuropsychiatric Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mickey BJ, White AT, Arp AM, Leonardi K, Torres MM, Larson AL, Odell DH, Whittingham SA, Beck MM, Jessop JE, Sakata DJ, Bushnell LA, Pierson MD, Solzbacher D, Kendrick EJ, Weeks HR 3rd, Light AR, Light KC, Tadler SC. Propofol for Treatment-Resistant Depression: A Pilot Study. Int J Neuropsychopharmacol. 2018 Dec 1;21(12):1079-1089. doi: 10.1093/ijnp/pyy085. PMID 30260415

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02935647/Prot_SAP_000.pdf